CLINICAL TRIAL: NCT05071105
Title: Stereotactic Ablative Body Radiotherapy in Elderly Women With Early Breast Cancer Unsuitable for Surgery and Elected to Receive Primary Endocrine Therapy Alone
Brief Title: SBRT in Early Breast Cancer in Elderly Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Laura Cedrone, Resident, University of Rome Tor Vergata
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 222.20
Record Dates: First submitted 2021-05-10; First posted 2021-10-07 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-12

CONDITIONS: Breast Neoplasm Female
Keywords: Radiotherapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Time to Event Key-Board, a dose escalation design study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 40Gy/5fx (Experimental): The starting dose level will be 8Gy x 5 fractions, i.e., 40 Gy/5 nonconsecutive once-daily fractions.
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- 42.5Gy/5fx (Experimental): The intermediate dose level will be 8.5Gy x 5 fractions, i.e. 42.5Gy/5 nonconsecutive once-daily fractions.
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- 45Gy/5fx (Experimental): The higher dose level will be 9Gy x 5 fractions, i.e. 45Gy/5 nonconsecutive once-daily fractions
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — In every group, the dose is prescribed at the edge of the PTV. To be approved, 95% of the PTV will be conformally covered by the prescription isodose surface and 99% of PTV will receive a minimum of 90% of the prescription dose.
  Other Names: SBRT; Stereotaxis; Stereotactic Radiotherapy

SUMMARY:
Surgical treatment represents the standard of local therapy in patients with early breast cancer, however in women over75, the comorbidities related to aging reduce the possibility of candidates for surgical treatment. In the United Kingdom it is estimated that over 40% of elderly women do not receive surgery for their breast cancer, and that their primary treatment is hormonal only, the so-called primary endocrinotherapy.

In Italy the recent AIOM guidelines of 2019 exclude, in patients with hormone-sensitive disease and age older than 70, the omission of surgery in favor of hormone therapy alone, thus underlining the importance of a treatment local. However, there are currently no local treatments that could in any way effectively control the primary tumor.

In recent years, SRT has widely found space as a therapeutic alternative in patients not fit for surgery.

Stereotactic Radiotherapy is a non-invasive treatment with ablative intent obtained with highly focused high intensity fields for a few fractions (generally 1-5). It is the standard treatment for surgically inoperable lung cancers, and is also used in the treatment of liver metastases, intermediate-risk prostate cancer and locally advanced pancreatic cancers. The applications of stereotactic treatment in breast cancer are limited to the neoadjuvant and adjuvant setting.

Against this backgroung, in elderly patients with localized breast cancer candidates for hormonal therapy and non-fit for surgery due to age or comorbidity, a SBRT could more effectively control local disease, not excluding local treatment rather than in itself it is considered very important.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer diagnosis in females; with population ageing, this diagnosis may increase in 75 years old or older patients.

According to AIRTUM data, 22% of new cases of breast cancer and 14% of death by breast cancer are expected in women over 70 years old.

Surgery is the gold standard of treatment for breast cancer, but advanced age and age-related comorbidity could reduce the ability of a surgical approach.

In the United Kingdom, it is estimated that over 40% of older women will not receive surgical treatment for breast tumor, while endocrine therapy alone is frequently offered. This treatment is known as primary endocrine therapy.

In our country, AIOM guidelines favor endocrine therapy alone in women over 70 with ER-positive tumors instead of surgical resection, even emphasizing the importance of local treatment.

Among nonsurgical methods to treat breast cancer, radiofrequency ablation and focused ultrasound have been investigated, but they are not widely available at present time.

Radiation therapy has been used to treat patients with inoperable breast cancer, but most of these treatments were palliative.

There are limited clinical data supporting the use of definitive conventionally fractionated radiotherapy and more specifically stereotactic ablative body radiotherapy in breast cancer.

A collaborative study between the Gustave-Roussy Institute and the Princess Margaret Hospital reviewed the use of radiotherapy alone as definitive breast cancer treatment.

Patients who had inoperable disease or who were unable to undergo general anesthesia received definitive hypofractionated radiotherapy (40Gy in 16 fractions, 45Gy in 20 fractions, or 45Gy in 18 fractions). This retrospective study demonstrated tumor dose as being a highly significant factor for local control, with very low rates of disabling complications at 10 years.

Van Limbergen et al. also performed a retrospective analysis of 221 patients withTis-T3N0-1 breast cancer treated with radiotherapy alone.

The risk of local recurrence was significantly associated with tumor size, age, radiation dose, and length of radiation. They concluded that doses needed to provide local control similar to a combination of surgery and radiation are 10 Gy higher for T1 tumors and 35Gy higher for T2 tumors.

Unfortunately, higher doses may result in worsened cosmetic outcomes. Van Limbergen et al reviewed 161 patients, and those that received dose higher than 75Gy recorded very poor cosmetic results in more than 30% of patients; if total dose was up to 80Gy only 15% of patients reported good cosmetic results.

It is important to remember that these papers are more than 25 years old, using older radiotherapy techniques and larger treatment fields.

With the development of modern radiation therapy techniques, and the adoption of Stereotactic Body RadioTherapy (SBRT) tumoricidal doses are delivered without severe complications.

SBRT is a non-invasive cancer treatment with ablative intent delivered with highly focused and accurate radiation beams for few fraction (generally 3-5 fractions).

Many trials established the safety and efficacy of SBRT in multiple organ sites including the lung, liver, spine, prostate and pancreas.

SBRT is actually shared as standard treatment in inoperable lung tumors: Timmerman et al. published one of the earlier extracranial SBRT trials on its use in early stage lung cancer, demonstrating excellent local control rates and side effect outcomes.

SBRT also offers a noninvasive alternative treatment for patients with liver metastases, who are not candidates for surgical resection.

The Stanford group initially established the safety of single fraction SBRT in 6 patients with locally advanced pancreatic cancer, subsequently a multi-institutional phase II study, reported by Herman et al. demonstrated equivalent efficacy in 1-year local progression freedom with acceptable toxicity profile in 49 patients with LAPC treated with 5 fractions SBRT following gemcitabine.

The scandinavian HYPO-RT-PC trial showed non-inferiority to conventionally fractionated radiotherapy for ultra-hypofractionated radiotherapy for intermediate-to-high risk prostate cancer regarding failure-free survival with similar late toxicity in both groups.

To date, SABR to primary tumor in breast cancer treatment has been mainly investigated in neoadjuvant and adjuvant setting. Bondiau et al. conducted a Phase I study involving 25 patients to determine the maximum tolerable dose of SBRT concomitant with neoadjuvant chemotherapy before surgery. Thirty-six percent of patients had a pathological complete response, with the highest rate (67%) at dose level of 25.5 Gy in 3 consecutive fractions. However, the maximum tolerated dose was not reached (highest dose level 31.5 in 3 consecutive fractions) as the group found that early SABR related toxicities were rare. Also in other studies toxicity was limited.

The first SBRT studies in the management of early stage breast cancer were post-operative studies. SBRT was used either as a boost, or for accelerated partial breast radiation therapy. Age was not an exclusion criterion, but mean ages were under 65 years. The proportion of patients aged >65 years were not given. SBRT has not yet been studied specifically in elderly patients who paradoxically most often have tumors with better histoprognostic factors than younger women.

Instead, SBRT role as a definitive ablative therapy in breast cancer is less considered and there are no prospective studies.

Therefore, in elderly patients (over 75y) eligible for hormone therapy only and unsuitable for surgery, SBRT could improve locoregional control by means of a short and highly effective treatment without any interruption of systemic treatment.

The Aim of this trial is to evaluate dose limiting toxicity for SBRT in elderly patients elected to receive hormone therapy only for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Histologically confirmed diagnosis of local disease only (cT1-T2 N0 M0)
* Luminal like A or B (estrogen receptor positive and/or progesterone receptor positive and Her2 negative Tumors)
* SBRT within 2 months after hormonal therapy start

Exclusion Criteria:

* Metastatic Disease
* Evidence of loco-regional nodal disease
* Multifocal or multicentric tumors
* Prior radiotherapy to the region of the study cancer that would result in overlap of therapy fields
* Concurrent systemic disorders that contraindicate radiotherapy

Min Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 6 months
  DLT is determined as any grade 3 or worse toxicity (per CTCAE v5.0) that occurs within 6 months from the start of SBRT

SECONDARY OUTCOMES:
Locoregional disease control (LRC) | 5 years
  Absence of progressive tumor within the radiation field, it also requires evidence of an objective response (50% reduction in the product of two dimensions of the dominant tumor mass for measurable disease, as per RECIST criteria)
Clinical complete response (cCR) | 6 months
  Disappearance of the target lesion; ideally, this determination will be made based on clinical evaluation and US and Rx Images
Cosmesis assesed by Harvard scale | 5 years
  Cosmesis evaluation will be carried out before treatment, at last day of treatment and at every clinical examination with Harris scale scoring system.
  The Harvard scale proposed by Harris et al., which has been used to evaluate cosmetic outcome after BCT, is a 4-point scale that describes the global esthetic appearance of breasts as excellent, good, fair, or poor.
Cosmesis assesed by BREAST-Q v2.0 | 5 years
  Cosmesis evaluation will be carried out before treatment, at last day of treatment and at every clinical examination with Breast-Q v2.0 questionnaire.
  The BREAST-Q v2.0 is a rigorously developed patient-reported outcome (PRO) measure designed to evaluate outcomes among women undergoing different types of breast treatment. Among the 6 BREAST-Q modules we will use "Physical well-being chest Module", "Satisfaction with breast Module" and "Adverse Effects of Radiation Module".
  All scales are transformed into scores that range from 0-100, a higher score means greater satisfaction or better QOL
Progression-free survival (PFS) | 5 years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.
Overall survival (OS) | 5 years
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
patient reported global health status assesed by EORTC QLC-C30 | 5 years
  Patient reported quality of life will be evaluated using the EORTC QLC-C30 v3.0 at time zero, at the end of treatment, at 6 and 12 months, and then yarly.
  The EORTC quality of life questionnaire (QLQ) is composed of both multi-item scales and single-item measures, which include functional scales, symptom scales, a QoL scale, and specific single items.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
patient reported therapy side effects assesed by EORTC QLQ-BR23 | 5 years
  Patient reported breast specific satisfaction will be evaluated using the EORTC QLQ-BR23 v3.0 at time zero, at the end of treatment, at 6 and 12 months, and then yarly.
  QLQ-BR23 is a supplementary questionnaire module for specific breast cancer populations; it incorporates 5 multi-item scales to assess systemic therapy side effects, arm and breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Maria D'Angelillo, Principal Investigator — Fondazione Policlinico Tor Vergata
Locations (1):
- Fondazione Policlinico Tor Vergata, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hind D, Wyld L, Beverley CB, Reed MW. Surgery versus primary endocrine therapy for operable primary breast cancer in elderly women (70 years plus). Cochrane Database Syst Rev. 2006 Jan 25;(1):CD004272. doi: 10.1002/14651858.CD004272.pub2. PMID 16437480
- [Background] Kinoshita T, Iwamoto E, Tsuda H, Seki K. Radiofrequency ablation as local therapy for early breast carcinomas. Breast Cancer. 2011 Jan;18(1):10-7. doi: 10.1007/s12282-009-0186-9. Epub 2010 Jan 14. PMID 20072824
- [Background] Schmitz AC, Gianfelice D, Daniel BL, Mali WP, van den Bosch MA. Image-guided focused ultrasound ablation of breast cancer: current status, challenges, and future directions. Eur Radiol. 2008 Jul;18(7):1431-41. doi: 10.1007/s00330-008-0906-0. Epub 2008 Mar 20. PMID 18351348
- [Background] Courdi A, Ortholan C, Hannoun-Levi JM, Ferrero JM, Largillier R, Balu-Maestro C, Chapellier C, Ettore F, Birtwisle-Peyrottes I. Long-term results of hypofractionated radiotherapy and hormonal therapy without surgery for breast cancer in elderly patients. Radiother Oncol. 2006 May;79(2):156-61. doi: 10.1016/j.radonc.2006.04.005. Epub 2006 May 15. PMID 16698099
- [Background] Arriagada R, Mouriesse H, Rezvani A, Sarrazin D, Clark RM, DeBoer G, Bush RS. Radiotherapy alone in breast cancer. Analysis of tumor and lymph node radiation doses and treatment-related complications. The experience of the Gustave-Roussy Institute and the Princess Margaret Hospital. Radiother Oncol. 1993 Apr;27(1):1-6. doi: 10.1016/0167-8140(93)90037-9. PMID 8327727
- [Background] Van Limbergen E, Van der Schueren E, Van den Bogaert W, Van Wing J. Local control of operable breast cancer after radiotherapy alone. Eur J Cancer. 1990;26(6):674-9. doi: 10.1016/0277-5379(90)90115-a. PMID 2168190
- [Background] Van Limbergen E, Rijnders A, van der Schueren E, Lerut T, Christiaens R. Cosmetic evaluation of breast conserving treatment for mammary cancer. 2. A quantitative analysis of the influence of radiation dose, fractionation schedules and surgical treatment techniques on cosmetic results. Radiother Oncol. 1989 Dec;16(4):253-67. doi: 10.1016/0167-8140(89)90037-6. PMID 2616812
- [Background] Timmerman R, Paulus R, Galvin J, Michalski J, Straube W, Bradley J, Fakiris A, Bezjak A, Videtic G, Johnstone D, Fowler J, Gore E, Choy H. Stereotactic body radiation therapy for inoperable early stage lung cancer. JAMA. 2010 Mar 17;303(11):1070-6. doi: 10.1001/jama.2010.261. PMID 20233825
- [Background] Schefter TE, Kavanagh BD, Timmerman RD, Cardenes HR, Baron A, Gaspar LE. A phase I trial of stereotactic body radiation therapy (SBRT) for liver metastases. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1371-8. doi: 10.1016/j.ijrobp.2005.01.002. PMID 16029795
- [Background] Herfarth KK, Debus J, Lohr F, Bahner ML, Rhein B, Fritz P, Hoss A, Schlegel W, Wannenmacher MF. Stereotactic single-dose radiation therapy of liver tumors: results of a phase I/II trial. J Clin Oncol. 2001 Jan 1;19(1):164-70. doi: 10.1200/JCO.2001.19.1.164. PMID 11134209
- [Background] Koong AC, Le QT, Ho A, Fong B, Fisher G, Cho C, Ford J, Poen J, Gibbs IC, Mehta VK, Kee S, Trueblood W, Yang G, Bastidas JA. Phase I study of stereotactic radiosurgery in patients with locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2004 Mar 15;58(4):1017-21. doi: 10.1016/j.ijrobp.2003.11.004. PMID 15001240
- [Background] Herman JM, Chang DT, Goodman KA, Dholakia AS, Raman SP, Hacker-Prietz A, Iacobuzio-Donahue CA, Griffith ME, Pawlik TM, Pai JS, O'Reilly E, Fisher GA, Wild AT, Rosati LM, Zheng L, Wolfgang CL, Laheru DA, Columbo LA, Sugar EA, Koong AC. Phase 2 multi-institutional trial evaluating gemcitabine and stereotactic body radiotherapy for patients with locally advanced unresectable pancreatic adenocarcinoma. Cancer. 2015 Apr 1;121(7):1128-37. doi: 10.1002/cncr.29161. Epub 2014 Dec 23. PMID 25538019
- [Background] Widmark A, Gunnlaugsson A, Beckman L, Thellenberg-Karlsson C, Hoyer M, Lagerlund M, Kindblom J, Ginman C, Johansson B, Bjornlinger K, Seke M, Agrup M, Fransson P, Tavelin B, Norman D, Zackrisson B, Anderson H, Kjellen E, Franzen L, Nilsson P. Ultra-hypofractionated versus conventionally fractionated radiotherapy for prostate cancer: 5-year outcomes of the HYPO-RT-PC randomised, non-inferiority, phase 3 trial. Lancet. 2019 Aug 3;394(10196):385-395. doi: 10.1016/S0140-6736(19)31131-6. Epub 2019 Jun 18. PMID 31227373
- [Background] Bondiau PY, Courdi A, Bahadoran P, Chamorey E, Queille-Roussel C, Lallement M, Birtwisle-Peyrottes I, Chapellier C, Pacquelet-Cheli S, Ferrero JM. Phase 1 clinical trial of stereotactic body radiation therapy concomitant with neoadjuvant chemotherapy for breast cancer. Int J Radiat Oncol Biol Phys. 2013 Apr 1;85(5):1193-9. doi: 10.1016/j.ijrobp.2012.10.034. Epub 2013 Jan 16. PMID 23332384
- [Background] Guidolin K, Yaremko B, Lynn K, Gaede S, Kornecki A, Muscedere G, BenNachum I, Shmuilovich O, Mouawad M, Yu E, Sexton T, Gelman N, Moiseenko V, Brackstone M, Lock M. Stereotactic image-guided neoadjuvant ablative single-dose radiation, then lumpectomy, for early breast cancer: the SIGNAL prospective single-arm trial of single-dose radiation therapy. Curr Oncol. 2019 Jun;26(3):e334-e340. doi: 10.3747/co.26.4479. Epub 2019 Jun 1. PMID 31285677
- [Background] Rahimi A, Thomas K, Spangler A, Rao R, Leitch M, Wooldridge R, Rivers A, Seiler S, Albuquerque K, Stevenson S, Goudreau S, Garwood D, Haley B, Euhus D, Heinzerling J, Ding C, Gao A, Ahn C, Timmerman R. Preliminary Results of a Phase 1 Dose-Escalation Trial for Early-Stage Breast Cancer Using 5-Fraction Stereotactic Body Radiation Therapy for Partial-Breast Irradiation. Int J Radiat Oncol Biol Phys. 2017 May 1;98(1):196-205.e2. doi: 10.1016/j.ijrobp.2017.01.020. Epub 2017 Jan 12. PMID 28586960
- [Background] van der Leij F, Bosma SC, van de Vijver MJ, Wesseling J, Vreeswijk S, Rivera S, Bourgier C, Garbay JR, Foukakis T, Lekberg T, van den Bongard DH, van Vliet-Vroegindeweij C, Bartelink H, Rutgers EJ, Elkhuizen PH. First results of the preoperative accelerated partial breast irradiation (PAPBI) trial. Radiother Oncol. 2015 Mar;114(3):322-7. doi: 10.1016/j.radonc.2015.02.002. Epub 2015 Feb 17. PMID 25701298
- [Background] Bondiau PY, Gal J, Chapellier C, Haudebourg J, Courdi A, Levy J, Gerard A, Sumodhee S, Maurin M, Chateau Y, Barranger E, Ferrero JM, Thariat J. Robotic Stereotactic Boost in Early Breast Cancer, a Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2019 Feb 1;103(2):374-380. doi: 10.1016/j.ijrobp.2018.09.020. Epub 2018 Oct 26. PMID 30612961
- [Background] Vermeulen S, Cotrutz C, Morris A, Meier R, Buchanan C, Dawson P, Porter B. Accelerated Partial Breast Irradiation: Using the CyberKnife as the Radiation Delivery Platform in the Treatment of Early Breast Cancer. Front Oncol. 2011 Nov 21;1:43. doi: 10.3389/fonc.2011.00043. eCollection 2011. PMID 22649764
- [Background] Lozza L, Fariselli L, Sandri M, Rampa M, Pinzi V, De Santis MC, Franceschini M, Trecate G, Maugeri I, Fumagalli L, Bonfantini F, Bianchi G, Pignoli E, De Martin E, Agresti R. Partial breast irradiation with CyberKnife after breast conserving surgery: a pilot study in early breast cancer. Radiat Oncol. 2018 Mar 23;13(1):49. doi: 10.1186/s13014-018-0991-4. PMID 29566762
- [Background] Obayomi-Davies O, Kole TP, Oppong B, Rudra S, Makariou EV, Campbell LD, Anjum HM, Collins SP, Unger K, Willey S, Tousimis E, Collins BT. Stereotactic Accelerated Partial Breast Irradiation for Early-Stage Breast Cancer: Rationale, Feasibility, and Early Experience Using the CyberKnife Radiosurgery Delivery Platform. Front Oncol. 2016 May 23;6:129. doi: 10.3389/fonc.2016.00129. eCollection 2016. PMID 27242967
- [Background] Livi L, Meattini I, Marrazzo L, Simontacchi G, Pallotta S, Saieva C, Paiar F, Scotti V, De Luca Cardillo C, Bastiani P, Orzalesi L, Casella D, Sanchez L, Nori J, Fambrini M, Bianchi S. Accelerated partial breast irradiation using intensity-modulated radiotherapy versus whole breast irradiation: 5-year survival analysis of a phase 3 randomised controlled trial. Eur J Cancer. 2015 Mar;51(4):451-463. doi: 10.1016/j.ejca.2014.12.013. Epub 2015 Jan 17. PMID 25605582
- [Background] Rahimi A, Zhang Y, Kim DW, Morgan H, Hossain F, Leitch M, Wooldridge R, Seiler S, Goudreau S, Haley B, Rao R, Rivers A, Spangler A, Ahn C, Stevenson S, Staley J, Albuquerque K, Ding C, Gu X, Zhao B, Timmerman R. Risk Factors for Fat Necrosis After Stereotactic Partial Breast Irradiation for Early-Stage Breast Cancer in a Phase 1 Clinical Trial. Int J Radiat Oncol Biol Phys. 2020 Nov 1;108(3):697-706. doi: 10.1016/j.ijrobp.2020.05.025. Epub 2020 May 26. PMID 32464155
- [Background] Murray Brunt A, Haviland JS, Wheatley DA, Sydenham MA, Alhasso A, Bloomfield DJ, Chan C, Churn M, Cleator S, Coles CE, Goodman A, Harnett A, Hopwood P, Kirby AM, Kirwan CC, Morris C, Nabi Z, Sawyer E, Somaiah N, Stones L, Syndikus I, Bliss JM, Yarnold JR; FAST-Forward Trial Management Group. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial. Lancet. 2020 May 23;395(10237):1613-1626. doi: 10.1016/S0140-6736(20)30932-6. Epub 2020 Apr 28. PMID 32580883
- [Background] Harris JR, Levene MB, Svensson G, Hellman S. Analysis of cosmetic results following primary radiation therapy for stages I and II carcinoma of the breast. Int J Radiat Oncol Biol Phys. 1979 Feb;5(2):257-61. doi: 10.1016/0360-3016(79)90729-6. No abstract available. PMID 110740
- See also: Related Info — http://www.aiom.it/i-numeri-del-cancro-in-italia/